CLINICAL TRIAL: NCT02877173
Title: Efficacy and Safety of Alprostadil Liposomes for Injection in the Treatment of Atherosclerotic Occlusive Disease of the Lower Extremities-A Phase II Multi-center Randomised Controlled Trial
Brief Title: A Safety/Efficacy Study of Alprostadil Liposomes for Injection to Treat Lower Extremity Arteriosclerosis Obliterans
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou Yipinhong Pharmaceutical CO.,LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YPH-ZZTP-L01
Record Dates: First submitted 2016-08-16; First posted 2016-08-24 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: Arteriosclerosis Obliterans
Keywords: Arteriosclerosis Obliterans; Atherosclerotic Occlusive Disease of the Lower Extremities; Intermittent Claudication
MeSH Terms: conditions — Arteriosclerosis Obliterans; Intermittent Claudication | interventions — Injections; Alprostadil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Alprostadil Liposomes for Injection (Experimental): Alprostadil Liposomes for Injection at low dose:20ug,once a day,continuous administration for 3 weeks; Alprostadil Liposomes for Injection at medium dose:40ug,once a day,continuous administration for 3 weeks; Alprostadil Liposomes for Injection at high dose:60ug,once a day,continuous administration for 3 weeks;
  Interventions: Drug: Alprostadil Liposomes for Injection
- Alprostadil Injection (Active Comparator): Alprostadil Injection:10ug,once a day,continuous administration for 3 weeks;
  Interventions: Drug: Alprostadil Injection

INTERVENTIONS:
Drug: Alprostadil Liposomes for Injection — 3 doses of Alprostadil Liposomes for Injection are 20ug/q.d,40ug/q.d,60ug/q.d.All groups will be continuous administration for 3 weeks.
  Other Names: No other names
  Arms: Alprostadil Liposomes for Injection
Drug: Alprostadil Injection — Alprostadil Injection(the positive control group):10ug/q.d,continuous administration for 3 weeks.
  Other Names: No other names
  Arms: Alprostadil Injection

SUMMARY:
A phase II,randomized,double-blind,multi-doses,positive drug parallel controlled,multi-center clinical trial to evaluate initially the efficacy and safety of alprostadil liposomes for injection in the treatment of atherosclerotic occlusive disease of the lower extremities.

DETAILED DESCRIPTION:
This is a phase 2 dose-finding study evaluating initially the efficacy and safety of alprostadil liposomes for injection in the treatment of atherosclerotic occlusive disease of the lower extremities at different dose strengths.The total duration of subject participation will be approximately 5 weeks,consisting of a 2-week run-in period,3-week treatment and safety follow-up period.

Subjects will sign the informed consent form(ICF) at a screening visit and will be assigned a subject identifier.Subjects meeting all inclusion/exclusion criteria and who have successfully completed all protocol procedures at screening will enter the 2-week run-in.Following the 2-week run-in period,eligible subjects will be randomized(1:1:1:1) to one of the following double-blind treatment groups:

Group A : Alprostadil Liposomes for Injection at low dose:20ug,once a day(QD); Group B : Alprostadil Liposomes for Injection at medium dose:40ug,QD Group C : Alprostadil Liposomes for Injection at high dose:60ug,QD Group D(Positive Control Group) : Alprostadil Injection:10ug,QD All treatments will be delivered by intravenously guttae.A subject will be consider to have completed the study when they have completed all phase of the study including run-in,randomization,the randomized treatment and efficacy and safety follow-up phase.

ELIGIBILITY:
Inclusion Criteria:

* An established clinical history of Atherosclerotic Occlusive Disease of the Lower Extremities in accordance with the definition by Chinese Medical Association(2015).
* Age>40
* Atherosclerotic Occlusive Disease of the Lower Extremities diagnosis
* Arterial ischemia of the lower extremities pulsation has been weakened or disappeared.
* Ankle brachial index(ABI) less than or equal to 0.9
* Diagnosis of artery stenosis or occlusion with imaging tests,including Doppler ultrasonography,CT angiogram(CTA),magnetic resonance angiography (MRA) or digital subtraction angiography(DSA) within 1 month prior to Screening.
* Fontaine stage classification:Stage II
* Distance of asymptomatic disease and claudication between 50m to 800m(The treadmill setting:pace at 3 km/h,incline at 12%).Subjects have intermittent claudication twice within 1 week prior to enrollment visit(Baseline is defined as the first measurement.Change from baseline in P-values less than or equal to 25%).
* Age:80 years old or younger.
* Intermittent claudication has been in stable condition in the last 6 months.And there was no history of exacerbations within 3 months prior to enrollment visit.
* Informed Consent:A signed and dated written informed consent prior to study participation.

Exclusion Criteria:

* Subjects who have cardiac disease including caradiac failure,arrhythmias,coronary disease,mitral or aortic stenosis.Subjects with a recent history of myocardial infarction within the past 6 months are to be excluded.
* Subjects who have pneumonedema,pulmonary infiltrates,interstitial pneumonia,severe chronic obstructive airway disorders or respiratory insufficiency confirmed by clinical examination.
* Liver:Subjects with abnormal liver function tests defined as aspartate aminotransferase(AST) or alanine aminotransferase(ALT) greater than equal to 1.5 times upper limit of normal,as well as a diagnosis of primary liver disease will be excluded.
* Renal:Subjects with abnormal kidney function tests defined as Creatinine clearance rate(SCr) greater than or equal to upper limit of normal.
* Clinically Uncontrolled Hypertension:Subjects who have clinically significant uncontrolled hypertension(Systolic blood pressure:greater than or equal to 180mmHg;Or diastolic blood pressure:greater than or equal to 110mmHg).
* Ankle systolic pressure is less than or equal to 50mmHg.
* Subjects with affected limbs surgery or endovascular treatment within 3 months prior to Screening.Subjects who received Prostanoids within the past 1 week are to be excluded.
* Subjects who received walking rehabilitation training successfully within the past 6 months.
* Subjects with a diagnosis of other diseases such as lower limb joint disorder,spinal lesions,neuropathy,serious lung and heart conditions which may impact intermittent claudication will be excluded.
* Subjects who have inflammation of the vascular disease including Takayasu's arteritis,edema perivascular.
* Subjects with active peptic ulcerease or bleeding tendency will be excluded.
* Glaucoma:Subjects with a diagnosis of glaucoma or high intraocular pressure will be excluded.
* Subjects who are medically unable to withhold their vasodilator including naftidrofuryl,pentoxy,buflomedil or cilostazol will be excluded.
* Subjects who received any powerful analgesic within 1 month perior to Screening.
* Subjects with a history of psychiatric disease or Alzheimer's Disease.
* Cancer:Subjects with a diagnosis of cancer will be excluded.
* Drug Allergy:Subjects who have a history of any componet of Alprostadil Injection.
* Previous Participation:Subjects who were previously enrolled in any clinical trial within 1 month period to Screening.
* Pregnancy:Women who are pregnant or lactating or women of childbearing potential who are not using an acceptable method of contraception.
* Subjects,who in the opinion of the Investigator,will not be fit for this study.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-07 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in distance of asymptomatic disease and claudication after 3 weeks of treatment. | After 3 weeks of treatment
  Unit of distance of asymptomatic disease and claudication:meters

SECONDARY OUTCOMES:
Change from baseline in maximun distance of claudication after 3 weeks of treatment. | After 3 weeks of treatment
  Unit of maximun distance of claudication :meters
Change from baseline in distance of asymptomatic disease and claudication and in maximum distance of claudication after 2 weeks of treatment. | After 2 weeks of treatment
  Unit of distance of asymptomatic disease and claudication:meters
The proportion of patients to treatment failure. | After 3 weeks of treatment
  The treatment failure is defined as arteriosclerosis obliterans(ASO) exacerbation that has necessary to change chemotherapy or have interventional operation.
Incidence of Adverse Events(AEs) | over 3 weeks of treatment
  The safety endpoints for this study include:
  1. AEs
  2. Vital Sign Measurements
  3. Physical examination
  4. Clinical Laboratory Evaluations

CONTACTS AND LOCATIONS:
Overall Officials: Yongquan Gu, Study Chair — Xuanwu Hospital, Beijing; Xiangchen Dai, Principal Investigator — Tianjing Medical University General Hospital; Bonan Lv, Principal Investigator — Hebei General Hospital; Jun Zhao, Principal Investigator — Shanghai Sixth People Hospital; Jichun Zhao, Principal Investigator — West China Hospital; Dan Liu, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University; Haofu Wang, Principal Investigator — The Affiliated Hospital of Qingdao University; Gang Zhao, Principal Investigator — First Affiliated Hospital of Heilongjiang Chinese Medicine University; Weiguang Guo, Principal Investigator — Second Affiliated Hospital of Heilongjiang University of Chinese Medicine; Qi Wang, Principal Investigator — The First Hospital of Jilin University; Xiwei Zhang, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Xuanwu Hospital Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No